CLINICAL TRIAL: NCT01381965
Title: Foveal Cone Outer Segment Resumption to Predict Visual Recovery After Macular Hole Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Kyorineye006; KYORIN-H21012 (Other: Kyorin University)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Macular Holes
Keywords: spectral-domain optical coherence tomography; idiopathic macular hole; cone outer segment tips line; vitrectomy
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eyes with macular hole (Active Comparator)
  Interventions: Procedure: Vitreous surgery for macular hole

INTERVENTIONS:
Procedure: Vitreous surgery for macular hole — Vitreous surgery for macular hole

SUMMARY:
Spectral domain optical coherence tomography (SD-OCT) was used to determine whether the repair of photoreceptor cone outer segment tips defect is significantly correlated with the visual outcomes after macular hole surgery.

DETAILED DESCRIPTION:
Spectral domain optical coherence tomography (SD-OCT) was used to calculate the mean length of photoreceptor cone outer segment tips (COST) defect on 1, 3, 6, 9, and 12 months after macular hole surgery. The correlation between the mean length of COST defect and the BCVA was determined. Prognostic factors might have influenced for COST repair was also evaluated by multivariable analysis.

ELIGIBILITY:
Inclusion Criteria:

* macular hole patients with surgically-closed hole

Exclusion Criteria:

* macular hole patients failed to close hole
* presence of retinal diseases including a treated rhegmatogenous retinal detachment, diabetic retinopathy, and high myopia with an axial length >27.0mm or refractive error > -8.0 diopters(D).
* patients who were not followed at least 6 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | one year
  Preoperative, postoperative 1, 3, 6, 9, 12 months

SECONDARY OUTCOMES:
Integrity of cone outer segment tips line | one year
  The mean length of cone outer segment tips defect on preoperative and postoperative 1, 3, 6, 9, and 12 months with spectral domain optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Makoto Inoue, Mitaka, Tokyo, Japan